CLINICAL TRIAL: NCT00863993
Title: Energy Expenditure and Gastric Bypass Surgery
Status: Withdrawn | Type: Observational
Why Stopped: no patients enrolled.
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, James Levine, Professor of Medicine, Mayo Clinic
Other Study IDs: 05-004359; R01DK072479 (NIH)
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Gastric Bypass Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study is to assess whether activity thermogenesis increases in patients undergoing bariatric surgery post-operatively compared to pre-operatively. The investigators will assess non-exercise activity thermogenesis using a validated Physical Activity Monitoring System and doubly labeled water, immediately pre-operatively and again at 6 and 18 months post-operatively. PAMS has been validated in lean and obese individuals. This is to assess energy expenditure, activity thermogenesis and NEAT during the phase of greatest weight loss and once weight loss has plateaued. This will permit us to address our primary hypothesis that activity thermogenesis as a fraction of total daily energy expenditure increases in patients undergoing bariatric surgery 6 and 18 months post-operatively, compared to pre-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing gastric bypass surgery, 18-60 years

Exclusion Criteria:

* Eligible subjects will be excluded who cannot walk at 2.4 mph for 15 minutes, or weigh greater than 227 kg at the screening visit.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 40 healthy patients (M=F, aged 18-60 years) undergoing gastric bypass bariatric surgery will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
TDEE (total daily energy expenditure) | March 2009 to October 2013
  Activity thermogenesis as a fraction of total daily energy expenditure increases in patients undergoing bariatric surgery 6 and 18 months post-operatively, compared to pre-operatively.